CLINICAL TRIAL: NCT01109459
Title: Multimodal Physician Intervention to Detect Amblyopia (Recruiting Title "Equipping Primary Care Physicians to Improve Care for Children")
Brief Title: Multimodal Physician Intervention to Detect Amblyopia
Acronym: EPPICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Wendy L. Marsh-Tootle, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: EY015893
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Amblyopia; Strabismus
Keywords: preschool; screening; cluster randomized; physician practice patterns; behavior; knowledge; attitudes; guideline adherence
MeSH Terms: conditions — Amblyopia; Strabismus; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pediatric vision screening (Experimental): intervention
  Interventions: Other: Pediatric vision screening
- Pediatric blood pressure screening (Active Comparator): control
  Interventions: Other: Pediatric blood pressure screening
- Primary care providers observation only (No Intervention): Observational

INTERVENTIONS:
Other: Pediatric blood pressure screening — Website presenting case-based education with tailoring based on knowledge and interactive with responses collected on line. Has a tool box for office materials to promote and encourage guideline based performance.
  Arms: Pediatric blood pressure screening
Other: Pediatric vision screening — Website presenting case-based education about amblyopia and strabismus with tailoring based on knowledge and interactive with responses collected on line. Has a tool box for office materials to promote and encourage guideline based performance.
  Arms: Pediatric vision screening

SUMMARY:
Current research shows low rates of quantitative vision screening at preschool ages in the medical home. This study targets providers (PCPs) to evaluate the effectiveness of a web-based intervention to improve knowledge about strabismus, amblyopia and preschool vision screening, to increase preschool vision screening rates, and to improve rates of diagnosis of strabismus and amblyopia by eye specialists.

DETAILED DESCRIPTION:
Despite decades of research showing adverse neural consequences of abnormal vision, little has changed for amblyopic children. Over the past 40 years, data have shown that most children with amblyopia are detected late. In our health care system, primary care physicians play a pivotal role in translating findings about amblyopia into practice. But, our experience with the Maternal and Child Health Bureau (MCHB) / NEI expert panel on Vision Screening in the Preschool Child and the MCHB/ American Academy of Pediatrics (AAP) Project Universal Preschool Vision Screening revealed that primary care physicians get very little training about amblyopia and risk factors. Consequently, many do not screen aggressively for these conditions.

The University of Alabama Departments of Optometry, Pediatrics and Continuing Medical Education, in collaboration Medicaid Agencies in Alabama, South Carolina and Illinois, have developed a novel, internet-based, multi-modal strategy to increase the understanding and recognition of amblyopia and its risk factors by pediatricians and primary care physicians in office based settings. We have designed a cluster-randomized, controlled clinical trial to test whether our intervention results in improved performance by "intervention" physicians compared to control physicians (exposed to a web-based intervention for pediatric blood pressure screening and adolescent chlamydia screening). Our design, along with pre / post-intervention and control / intervention performance measures, will evaluate changes in practice attributable to the intervention versus those occurring from other sources over time. Our final analysis will show whether preschool patients of intervention physicians are more likely to be identified with strabismus or amblyopia. This research forges a critical link between the truly phenomenal body of amblyopia research fostered by the NEI and the health care offered to American children.

ELIGIBILITY:
Inclusion Criteria:

* files Medicaid claims for at least 8 well child visits for children aged 3 or 4 years during one year,
* files claims under individual name,
* has internet access.

Exclusion Criteria:

* files fewer than 8 Medicaid claims for well child visits for children aged 3 or 4 years old during one year,
* files claims under a clinic name,
* does not have internet access.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2004-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
preschool vision screening by primary care providers | 1 year
  A rate: number of claims for preschool vision screening (using a billing procedure code) / number of claims for well child exams (another billng code). These procedure codes are filed by primary care providers (PCPs). Rates are determined for individual Intervention, Control and non-participating eligible PCPs.

SECONDARY OUTCOMES:
Diagnosis of strabismus or amblyopia by eye specialists | 1 year
  A rate: number of claims from eye specialists with procedure codes of strabismus or amblyopia(using billing data) / number of claims for well child exams by intervention, control and non-participating eligible PCPs.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Marsh-Tootle, OD,MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Marsh-Tootle WL, Frazier MG, Kohler CL, Dillard CM, Davis K, Schoenberger YM, Wall TC. Exploring pre-school vision screening in primary care offices in Alabama. Optom Vis Sci. 2012 Oct;89(10):1521-31. doi: 10.1097/OPX.0b013e318269ca9f. PMID 22982768
- [Derived] Marsh-Tootle WL, McGwin G, Kohler CL, Kristofco RE, Datla RV, Wall TC. Efficacy of a web-based intervention to improve and sustain knowledge and screening for amblyopia in primary care settings. Invest Ophthalmol Vis Sci. 2011 Sep 9;52(10):7160-7. doi: 10.1167/iovs.10-6566. PMID 21730344
- [Derived] Wall TC, Marsh-Tootle WL, Crenshaw K, Person SD, Datla R, Kristofco RE, Hartmann EE. Design of a randomized clinical trial to improve rates of amblyopia detection in preschool aged children in primary care settings. Contemp Clin Trials. 2011 Mar;32(2):204-14. doi: 10.1016/j.cct.2010.10.009. Epub 2010 Oct 23. PMID 20974292